CLINICAL TRIAL: NCT03046940
Title: The Influence of Doctor-patient Communication on Patients' Willingness to Take Medication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Winfried Rief, Professor, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016-37v-r
Record Dates: First submitted 2017-01-30; First posted 2017-02-08 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): No communication with a doctor
- Patient-centered (Experimental): Participants communicate with a doctor that uses a patient-centered style of communication
  Interventions: Other: Patient-centered style of communication
- Doctor-centered (Experimental): Participants communicate with a doctor that uses a doctor-centered style of communication
  Interventions: Other: Doctor-centered style of communication

INTERVENTIONS:
Other: Patient-centered style of communication — Different doctor-patient communication
  Arms: Patient-centered
Other: Doctor-centered style of communication — Different doctor-patient communication
  Arms: Doctor-centered

SUMMARY:
The experiment aims at investigating whether the doctor-patient communication has an influence on patients' willingness to take medication. Patients' attitude towards the medication is manipulated via a critical film sequence. Afterwards patients of the two experimental groups have a communication with one of the investigators of the study. Patients are told that the investigator is a medical doctor. The "doctors" either communicate in a patient-centered or doctor-centered style with the patient. Patients in the control group do not have the possibility to talk to a "medical doctor". Afterwards patients are offered the aforementioned pill that is supposed to be a cognitive enhancer (actually placebo pill). Pill intake is voluntary. The investigators hypothesize that patients in the experimental group with the patient-centered style of communication are more likely to take the pill than patients in the experimental group with the doctor-centered style of communication or patients in the control group.

ELIGIBILITY:
Inclusion Criteria:

* female
* between 18 and 35 years
* healthy
* adequate ability to see
* fluent in German (reading and writing)

Exclusion Criteria:

* regular intake of cognitive enhancers/medication that enhances concentration
* intake of psychotropic drugs
* medical or pharmacy students, advanced psychology students
* participants who know the investigators

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Pill intake | Within 10 minutes after doctor-patient communication
  Behavioural test

SECONDARY OUTCOMES:
Willingness to take medication (VAS) | Within 10 minutes prior to watching the film sequence, directly (within 5 minutes) after the film sequence, directly (within 10 minutes) after doctor-patient communication
  Visual analogue scale (VAS)
Critical attitude towards the medication (VAS) | Within 10 minutes prior to watching the film sequence, directly (within 5 minutes) after the film sequence, directly (within 10 minutes) after doctor-patient communication
  Visual analogue scale (VAS)
Influence on concentration (Concentration task) | Directly (within 10 minutes) after the pill was offered
  Concentration task

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, PhD, Prof, Principal Investigator — Philipps University Marburg
Locations (1):
- Department of Clinical Psychology and Psychotherapy, Philipps-University Marburg, Marburg, Germany